CLINICAL TRIAL: NCT03447392
Title: Discharge Education of Integrated Traditional and Western Medicine Reduces Re-hospitalization in Patients With Chronic Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Jguo
Record Dates: First submitted 2018-02-16; First posted 2018-02-27 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Heart Failure
Keywords: Patient Education; Chinese Medicine
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patient education and Chinese medicine (Experimental): 1-hour, one-on-one teaching session with a educator to the standard discharge education of Integrated Traditional and Western Medicine
  Interventions: Behavioral: Discharge Education of Chinese Medicine
- patient education (No Intervention): no discharge education

INTERVENTIONS:
Behavioral: Discharge Education of Chinese Medicine — Discharge Education of Integrated Traditional and Western Medicine
  Arms: patient education and Chinese medicine

SUMMARY:
Although interventions combining patient education and postdischarge management have demonstrated benefits in patients with chronic heart failure, the benefit attributable to patient education alone is not known. The investigators hypothesized that a patient discharge education program would improve clinical outcomes in patients with chronic heart failure.

DETAILED DESCRIPTION:
Although interventions combining patient education and postdischarge management have demonstrated benefits in patients with chronic heart failure, the benefit attributable to patient education of Integrated Traditional and Western Medicine is not known. The investigators hypothesized that a patient discharge education of Integrated Traditional and Western Medicine program would improve clinical outcomes in patients with chronic heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for this study were admitted to the hospital with a diagnosis of heart failure and documented left ventricular systolic dysfunction (ejection fraction<0.40).

Exclusion Criteria:

* CKD4 and CKD5

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2018-01-08 (Actual); Study Completion 2018-01-08 (Actual)

PRIMARY OUTCOMES:
total number of days hospitalized | 84 days
  total number of days hospitalized in the 84-day follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Xu ZOU, Study Chair — The Second Clinical College, Guangzhou University of Chinese Medicine
Locations (1):
- Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong, China